CLINICAL TRIAL: NCT02055287
Title: An Open-Label, Single Ascending Dose Pharmacokinetic and Safety Study of LY03004 Following Escalating Single Intramuscular Injection in Stable Patients With Schizophrenia or Schizoaffective Disorder
Brief Title: Pharmacokinetic and Safety Study of LY03004 in Stable Patients With Schizophrenia or Schizoaffective Disorder
Acronym: LY03004SAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY03004
Record Dates: First submitted 2014-01-31; First posted 2014-02-05 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY03004- 12.5 (Experimental): LY03004 dosage strength at 12.5mg
  Interventions: Drug: LY03004
- LY03004 - 25 (Experimental): LY03004 Dose Strength 25mg
  Interventions: Drug: LY03004
- LY03004- 37.5 (Experimental): LY03004 Dose Strength 37.5mg
  Interventions: Drug: LY03004
- LY03004 - 50 (Experimental): LY03004 Dose Strength 50mg
  Interventions: Drug: LY03004

INTERVENTIONS:
Drug: LY03004

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics (PK) of LY03004 following an escalating single intramuscular injection at 12.5, 25, 37.5, or 50 mg; and to evaluate the safety and tolerability and preliminary efficacy of LY03004 following intramuscular injection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 65 years old;
2. Patients must have a DSM-IV diagnosis of schizophrenia or schizoaffective disorder based on the Mini-International Neuropsychiatric Interview (MINI);
3. Patients must be clinically stable on antipsychotic medications other than risperidone or paliperidone or clozapine for at least 4 weeks prior to screening, based on clinical assessments and a Positive and Negative Syndrome Scale (PANSS) total score less than or equal to 70 at screening visit;
4. Patients with a Body Mass Index in range of 18.0 to 35.0;
5. Patients with an Informed consent form signed by the patient or legally acceptable representative

Exclusion Criteria:

1. Patients with a mental disorders other than schizophrenia or schizoaffective disorder, according to the DSM-IV;
2. Patients who received oral risperidone or paliperidone or clozapine within 14 days prior to screening, or Risperdal Consta within 100 days prior to screening or paliperidone palmitate within 10 months prior to screening;
3. Patients with neuroleptic malignant syndrome or physical fatigue associated with dehydration or malnutrition;
4. Patients who pose a significant risk of a suicide attempt based on history, investigator's judgment or have answered "yes" on the questions 4 or 5 for current or past 30 days on the screening form of the Columbia Suicide Severity Rating Scale (C-SSRS).
5. Patients with a history of sensitivity to akathisia and other EPS, especially with previous use of risperidone or paliperidone.
6. Patients with uncontrolled diabetes mellitus as indicated by a HbA1c level greater than or equal to 7%;
7. Patients with a history of or currently having epilepsy or convulsion disorders;
8. Patients who have had electroconvulsive therapy within the past 2 months prior to screening;
9. Patients who used medication known to be an inducer or inhibitor for CYP 2D6 less than 2 weeks prior to screening;
10. Patients with a history of allergic reaction to risperidone or to the excipients of LY03004;
11. Patients who have met DSM-IV-TR criteria for substance abuse or dependence with the exception of caffeine or nicotine in the past 6 months prior to screening
12. Patients with a history of clinically relevant cardiac arrhythmia's, cardiovascular disease, thyrotoxicosis, parkinsonism, or hemorrhagic diathesis;
13. Patients who are currently taking medications with primarily CNS activities such as antidepressants, mood stabilizers or anticonvulsants;
14. Patients who have participated in a clinical trial of another investigational drug within 30 days prior to screening;
15. Female patients who are pregnant or are breastfeeding or are of childbearing potential without adequate contraception.
16. Patients who have any clinically relevant hepatic, renal and cardiac dysfunction, or other medical condition or laboratory abnormality, which in the judgment of the investigator would interfere with the subject's ability to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Cmax for the Pharmacokinetics (PK) of LY03004 | 43 Days

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 43 Days
The change of the PANSS score for the Preliminary efficacy of LY03004 | 43 Days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Neuropsychiatric Research Center of Orange County, Orange, California
  - Community Clinical Research Inc, Austin, Texas

REFERENCES:
- [Derived] Wang W, Wang X, Dong Y, Walling DP, Liu P, Liu W, Shi Y, Sun K. Population Pharmacokinetic Analysis to Support and Facilitate Switching from Risperidone Formulations to Rykindo in Patients with Schizophrenia. Neurol Ther. 2024 Apr;13(2):355-372. doi: 10.1007/s40120-024-00578-w. Epub 2024 Jan 20. PMID 38244179